CLINICAL TRIAL: NCT01244178
Title: Hyperinsulinemic Therapy in Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: peter metrakos (Other)
Responsible Party: Sponsor-Investigator, peter metrakos, Associate Professor of Surgery and Associate Professor in Anatomy and Cell Biology McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 10-003-GEN
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Sepsis
Keywords: Sepsis; Insulin
MeSH Terms: conditions — Sepsis; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tight Glucose Control Hyperinsulinemic Group (Experimental)
  Interventions: Drug: Insulin
- Non-Tight Glucose Control Hyperinsulinemic Group (Experimental)
  Interventions: Drug: Insulin
- Standard Insulin Protocol Group (Active Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Intravenous Hyperinsulinemic therapy
  Arms: Non-Tight Glucose Control Hyperinsulinemic Group; Tight Glucose Control Hyperinsulinemic Group
Drug: Insulin — Standard Intravenous Insulin Therapy
  Arms: Standard Insulin Protocol Group

SUMMARY:
Insulin regulates blood sugar and acts to suppress inflammation. Hyperinsulinemic Therapy is a protocol for Insulin administration that involves the administration of a calculated higher dose of insulin into the blood stream. This therapy is called dextrose/insulin clamp. It has been shown to be safe and successful in maintaining normal glucose levels.

The objective of the study is to assess if the clamp can achieve a steady and normal blood glucose level in patients admitted to the intensive care unit with sepsis. Furthermore, if the higher insulin dose would lead to a drop in the inflammatory response seen in septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU with a diagnosis of Septic shock or Severe Sepsis.

Exclusion Criteria:

* Age less than 18 years old.
* Pregnancy.
* Patients who cannot provide informed consent and there is no surrogate decision maker.
* A delay of more than 24 hours between eligibility and randomization.
* Patients admitted to the intensive care unit for treatment of diabetic ketoacidosis or hyperosmolar state.
* Imminent death.
* Patients who the treating clinicians are not committed to full supportive care. This is confirmed by a documented treatment-limitation order that exceeds a "do-not-resuscitation" order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Glucose Control | During ICU stay (average one week)
  Measures glucose control using the hyperinsulinemic/normoglycemic clamp in patients with septic shock

SECONDARY OUTCOMES:
Inflammatory cytokines and biochemical hormonal response | At randomization then at 6,24, 120 hours
  Measurement of specific cytokines and hormonal responses to hyperinsulinemic therapy in patients with septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Peter Metrakos, FRCSC, Principal Investigator — McGill University
Locations (3):
- Canada (2):
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
- King Khalid Univesity Hospital, Riyadh, Riyadh Region, Saudi Arabia